CLINICAL TRIAL: NCT00196391
Title: A Multicenter Study to Evaluate Induction of Withdrawal Bleeding After Administration of DR-2021 in Women With Secondary Amenorrhea
Brief Title: A Trial to Evaluate DR-2021 in Women With Secondary Amenorrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Duramed Protocol Chair, Duramed Research, Inc.
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR-MPG-201
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-05

CONDITIONS: Amenorrhea
Keywords: secondary amenorrhea; progesterone
MeSH Terms: conditions — Amenorrhea | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental)
  Interventions: Drug: DR-2021a
- 2 (Experimental)
  Interventions: Drug: DR-2021b
- 3 (Experimental)
  Interventions: Drug: DR-2021c
- 4 (Experimental)
  Interventions: Drug: DR-2021d
- 5 (Experimental)
  Interventions: Drug: DR-2021e
- 6 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DR-2021a — 1 capsule daily for 10 days
  Other Names: Micronized progesterone
  Arms: 1
Drug: DR-2021b — 1 capsule daily for 10 days
  Other Names: Micronized Progesterone
  Arms: 2
Drug: DR-2021c — 1 capsule daily for 10 days
  Other Names: Micronized Progesterone
  Arms: 3
Drug: DR-2021d — 1 capsule daily for 10 days
  Other Names: Micronized Progesterone
  Arms: 4
Drug: DR-2021e — 1 capsule daily for 10 days
  Arms: 5
Other: Placebo — 1 matching placebo capsule for 10 days
  Arms: 6

SUMMARY:
This is a multicenter trial to compare the effectiveness of 4 doses of DR-2021 with placebo and oral micronized progesterone in inducing withdrawal bleeding in women with secondary amenorrhea.

DETAILED DESCRIPTION:
In this multicenter trial patients will be randomized to receive DR-2021, oral micronized progesterone, and placebo to evaluate the effects on withdrawal bleeding in women with secondary amenorrhea. Patients will be treated for 10 days and study participation will be approximately 24 days. Patients will undergo a physical exam including a pelvic and breast exam. Patients will be required to complete bleeding and spotting information daily in a diary.

ELIGIBILITY:
Inclusion Criteria:

* Not pregnant
* Secondary amenorrhea or oligomenorrhea of at least 50 days duration
* Not currently on any hormonal medication
* Not at risk of pregnancy or willing to use a non-hormonal method of birth control during the study (ie, condom)

Exclusion Criteria:

* Use an injectable or implantable estrogens, progestins, or androgens within the last 6 months
* Use of any hormonal birth control within the last 3 months
* Any contraindication to the use of progestins

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who have received 10 days of treatment and reported withdrawal bleeding. | Throughout study period

SECONDARY OUTCOMES:
Time to onset, duration, and severity of withdrawal bleeding. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Protocol Chair, Study Chair — Duramed Research, Inc.
Locations (25):
- United States (25):
  - Duramed Investigational Site, Mobile, Alabama
  - Duramed Investigational Site, Phoenix, Arizona
  - Duramed Investigational Site, Tucson, Arizona
  - Duramed Investigational Site, Carmichael, California
  - Duramed Investigational Site, San Diego, California
  - Duramed Investigational Site, Colorado Springs, Colorado
  - Duramed Investigational Site, Pueblo, Colorado
  - Duramed Investigational Site, Gainesville, Florida
  - Duramed Investigational Site, Leesburg, Florida
  - Duramed Investigational Site, Miami, Florida
  - Duramed Investigational Site, Atlanta, Georgia
  - Duramed Investigational Ste, Dawsonville, Georgia
  - Duramed Investigational Site, Douglasville, Georgia
  - Duramed Investigational Site, Laurel, Maryland
  - Duramed Investigational Site, St Louis, Missouri
  - Duramed Investigational Site, Alliance, Nebraska
  - Duramed Investigational Site, Lawrenceville, New Jersey
  - Duramed Investigational Site, Medford, Oregon
  - Duramed Investigational Site, Pittsburgh, Pennsylvania
  - Duramed Investigational Site, Willow Grove, Pennsylvania
  - Duramed Investigational Site, Columbia, South Carolina
  - Duramed Investigational Site, Memphis, Tennessee
  - Duramed Investigational Site, Dallas, Texas
  - Duramed Investigational Site, Houston, Texas
  - Duramed Investigational Site, Newport News, Virginia